CLINICAL TRIAL: NCT00974519
Title: Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Trials on the Effect of Combination of TCM and HAART on Immune Reconstitution of HIV/AIDS Patients
Brief Title: The Effect of Combination of Traditional Chinese Medicine (TCM) and Highly Active Antiretroviral Therapy (HAART) on Immune Reconstitution of HIV/AIDS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: WANG, Jie/Professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.07.16-2
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-09

CONDITIONS: Acquired Immune Deficiency Syndrome Virus; HIV Infections
Keywords: ADIS; complementary therapies
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fuzheng 3 (Active Comparator): Immunity 3 (Fuzheng 3), 8.75g / twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Interventions: Drug: Fuzheng 3
- Fuzheng 1 (Active Comparator): Immunity 1 (Fuzheng 1), 8.75g / twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Interventions: Drug: Fuzheng 1
- Placebo (Placebo Comparator): Placebo, 8.75g / twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fuzheng 3 — Immunity 3 (Fuzheng 3), 8.75g / twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Immunity 1 (Fuzheng 1) simulation agent, 8.75g / twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Arms: Fuzheng 3
Drug: Fuzheng 1 — Immunity 1 (Fuzheng 1), 8.75g / twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Immunity 3 (Fuzheng 3) simulation agent, 8.75g / twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Arms: Fuzheng 1
Drug: Placebo — Immunity 1 (Fuzheng 1) simulation agent, 8.75g / twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Immunity 3 (Fuzheng 3) simulation agent, 8.75g / twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Arms: Placebo

SUMMARY:
Immunity 1 (Fuzheng 1) is composed of herbs which have tonic and detoxific function. The long-term clinical application has proved the safety and effect. It can improve the symptoms and signs in AIDS patients with the effective rate of 70% and can significantly improve the quality of life. It can also improve and stabilize immune function and inhibit viral replication. The basis study have shown that Immunity 1 (Fuzheng 1) can inhibit viral replication from multi-target, multi-link, enhance immune function, increase the secretion of IL-2, IFN-γ, participate in immune regulation effect, enhance NK cell activity, promote CD3+CD4+T cell proliferation and increase macrophage phagocytes capacity.

DETAILED DESCRIPTION:
* Meng Kun found that Joint application of Chuankezhi can enhance the number of CD4 cells and reduce side-effects of HAART compared with HAART alone. in order to verify the long-term efficacy of combination therapy, they carried out an clinical observations of three cases of patients who received combination therapy for over a period of 3 years, through the observation of three cases of patients, they found that CD3+CD4+T lymphocyte count were significantly increased and HIV-RNA viral load were below 50copies for long-term, and without the occurrence of drug resistance. And the patient's symptoms and signs have also been significantly improved.
* Duan Cheng Yu analyses 334 cases of AIDS patients' clinical symptoms, signs and Karnofsky score, and CD3+CD4+ T lymphocyte count before and after treatment. The patients all take "kang ai bao sheng" capsules for 3 months. The results showed that 334 cases of patients receiving traditional Chinese and western medicine treatment shows improvement in symptoms and signs, increase in CD3+CD4+ T lymphocyte count. They proposed that combination of traditional Chinese and western medicine can improve symptoms, enhance immunity function and improve the quality of life of AIDS patients.
* In order to observe the effect of combination of TCM and HAART on HIV/AIDS patients, ZHANG Ai-min divided 63 cases of AIDS into 3 groups. 20 cases received TCM treatment and 22 cases received combination of TCM and HAART, 21 cases received western medicine. The patients' symptoms, signs, Karnofsky score points, CD3+CD4+T lymphocyte counts and HIV-RNA viral load were recorded and compare the difference between the 3 groups. The results showed that combination treatment can more effectively improve the immune function of HIV/AIDS patients, reduce HIV-RNA viral load, and improve the patients' symptoms, signs and the quality of life.
* Immunity 1 (Fuzheng 1) is composed of herbs which have tonic and detoxific function. The long-term clinical application has proved the safety and effect. It can improve the symptoms and signs in AIDS patients with the effective rate of 70% and can significantly improve the quality of life. It can also improve and stabilize immune function and inhibit viral replication. The basis study have shown that Immunity 1 (Fuzheng 1) can inhibit viral replication from multi-target, multi-link, enhance immune function, increase the secretion of IL-2, IFN-γ, participate in immune regulation effect, enhance NK cell activity, promote CD3+CD4+T cell proliferation and increase macrophage phagocytes capacity.
* Through the clinical trials, we are going to evaluate the efficacy and safety of combination of TCM and HAART on immune reconstitution of HIV/AIDS patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV antibody-positive, confirmed by Western Blot test
* CD 4 count ≤ 350 cells / ul
* Age ≥ 18 years old and ≤ 70 years old
* Voluntary participated in this study, signed informed consent form, and could be followed-up

Exclusion Criteria:

* Serious opportunistic infections were not brought under control (Pneumocystis carinii pneumonia, meningitis, esophageal candidiasis, lymphoma, toxoplasma encephalopathy, tuberculosis, etc.) before the experiment
* Participated in clinical trials of other drugs within one month before the experiment
* Received antiretroviral therapy or are anti-HIV drugs such as nucleoside reverse transcriptase inhibitors (NRTIs), non-nucleoside reverse transcriptase inhibitors (NNRTIs), protease inhibitors (PIs) and fusion-inhibiting agent (FIs), integrase inhibitors, inhibitors penetration within one month before the experiment
* Received immunomodulatory treatment within one month before the experiment WBC <2 × 10 9 / L, N <1.0 × 10 9 / L, Hb <90g / L, PLT <75 × 10 9 / L, liver and kidney dysfunction (AST, ALT, T-BIL ≥2 times of upper limit of the reference value or creatinine ≥ 2 times of the upper limit of reference value)
* Patients with pancreatitis or active gastric ulcer
* Patients with obvious active diseases in respiratory system, digestive system, circulatory system, blood system, neuroendocrine system, or genitourinary system diseases
* Persons suffering from autoimmune diseases
* Cancer patients which need chemotherapy
* Pregnant or lactating women, and did not use safe contraceptive measures for women of child-bearing age, as well as the male that can not take a reasonable method of contraception in trial period
* Hypersensitive people
* Patients with dysgnosia or language barriers, which can not fully understand the test or cooperate well

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood CD3+ CD4+ counts | 6 months

SECONDARY OUTCOMES:
Immune reconstitution efficiency | 6 months
Viral load | 6 months
Clinical symptoms and signs | 6 months
KPS score | 6 months
Quality of life score | 6 months
Side effect of HAART | 6 months
Safety evaluation | 6 months
Economic evaluation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jie WANG, MD, Study Chair — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Jie, WANG, Beijing, Beijing Municipality, China